CLINICAL TRIAL: NCT00508664
Title: Randomised Phase II Screening Study to be Used in an TP/TPF-chemotherapy (Short Induction) Before TP/TPF-induction, Radiotherapy With or Without Cetuximab in the Primary Therapy of the Only by Laryngectomy Operable Carcinoma of the Larynx/Hypopharynx
Brief Title: Docetaxel, Cisplatin (TP) + Radiation +/- Cetuximab in Larynx Carcinoma (CA)
Acronym: DeLOS II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ClinAssess (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Sanofi (Industry)
Responsible Party: Sponsor-Investigator, ClinAssess, Prof. Dietz, Universität Leipzig, University of Leipzig
Organization: University of Leipzig (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP(F)+Radiation+/-Cetuximab
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Squamous Cell Carcinoma of the Hypopharynx; Larynx Carcinoma
Keywords: by laryngectomy operable carcinoma of the larynx and the hypopharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms | interventions — Radiation; Cetuximab; Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): TP + Radiation (TPF until Feb 2009)
  Interventions: Radiation: Radiation; Drug: Docetaxel; Drug: Cisplatin (TP); Drug: 5-Fluorouracil (TPF) (only until Feb 2009)
- B (Experimental): TP + Cetuximab + Radiation (TPF until Feb 2009)
  Interventions: Radiation: Radiation; Drug: Cetuximab; Drug: Docetaxel; Drug: Cisplatin (TP); Drug: 5-Fluorouracil (TPF) (only until Feb 2009)

INTERVENTIONS:
Radiation: Radiation — Radiation start in week 11
Drug: Cetuximab — Day 1 400mg/m2 i.v. than weekly 250 mg/m2 i.v. for 16 weeks
  Arms: B
Drug: Docetaxel — 75 mg/m2 i.v. day 1 3 times
  Other Names: Taxotere
Drug: Cisplatin (TP) — 75 mg/m2 i.v. day 1 3 times
Drug: 5-Fluorouracil (TPF) (only until Feb 2009) — Only patients recruited until Feb 2009: 750 mg/m2 i.v. day 1-5, 3 times

SUMMARY:
The DeLOS II trial is a multicenter randomised phase II trial investigating a TP/5-Fluorouracil (TPF)-chemotherapy with or without cetuximab for Patients with only by laryngectomy operable carcinoma of the larynx/hypopharynx. Patients were divided in responder or non-responder after 4 weeks. Since August 2009 Responder receive TP with or without Cetuximab + radiation. (Until february 2009 Responder received TPF with or without Cetuximab + radiation.) Planned accrual is 85 patients per treatment arm. The primary study endpoint is a confirmatory proof of an adequate survival rate with a functionally larynx-conserving 2 years after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, primary only with laryngectomy respectable squamous-cell carcinoma of the larynx or hypopharynx
* T3-T4a carcinoma of the glottis
* T2-T4a carcinoma of the supraglottic, only controllable by laryngectomy and if applicable by root of tongue segmental resection
* T2-T4a carcinoma of the hypopharynx only controllable by laryngectomy (for example T2, post cricoidal) and hypopharynx segmental resection
* N-status: cervical metastases (N0-N3) have to be rehabilitate by surgical procedures

  * Blood count: Leukocytes >3500/mm\3, Neutrophils > 1500/ mm\3, Thrombocytes > 8000/ mm\3
  * Clinical chemistry:
* adequate renal function, defined by serum creatinine and urea not higher than 25% upper NL, creatinine-clearance > 60 ml/min/1,72 m\2
* adequate hepatic function with SGOT, SGPT not higher than 50% and bilirubin not higher than upper NL
* electrolytes at NL

  * anesthetic risk normal or low-grade elevated
  * age 18-75 years
  * written informed consent
  * effective contraception after individual advice for men and women if there is a possibility of reproductive potential (effective contraception are: oral contraception with estrogen and gestagen (no minipill), vaginal ring, contraception patch, estrogen free ovulation suppressors, hormone spiral with progesterone, injection for three month with depot gestagen, hormone releasing implantation (luteal hormone containing rod), abstinence or sterilization (vasectomy) of the male)

Exclusion Criteria:

* primary cancer treatable by operational larynx -conserving procedures
* distant metastases (M1-Status)
* total tumor volume exceeding 80 ml or larynx skeleton punctuated with infiltration of surrounding soft tissues respectively the esophageal aditus (exclusive cartilage infiltration represents no exclusion criteria)
* tumor-specific prior chemo or radiotherapy
* metachronous or synchronous malignant tumor (exception basalioma) [in case of a controlled tumor of different localization with a non-treated interval over 5 years to the present therapy the patient can be included after consultation with the coordinating investigator]
* life expectancy < 3 month
* Karnofsky performance status < 70%
* serious cardiopulmonary concomitant disease (cardiac insufficiency grade III and IV according NYHA status, myocardial infarction, angina pectoris, respiratory global insufficiency)
* Chronic diseases with permanent-therapy (uncontrolled diabetes, active rheumatoid arthritis)
* recurrent pneumonia, COPD GOLD stage <2, chronic inflammation of intestine or any other concomitant diseases, which disallow study participation in the opinion of the responsible physician
* Other circumstances (contra-indications), which disallow treatment with Docetaxel, Cisplatin, 5-FU, Cetuximab or radiotherapy
* Expected absent patient compliance
* Periodic follow-up not possible (for example address outside germany)
* Pregnant or breast-feeding woman
* Absent or constricted legal capacity
* Participation to another clinical trial with any investigational study within 30 days prior to study screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Confirmatory proof of an adequate survival rate with a functionally larynx-conserving 2 years after randomisation | LFS-rate 2 years after randomisation

SECONDARY OUTCOMES:
Descriptive analysis of the study arms concerning the secondary end criteria of the study | LSF 2 years after randomisation
Explorative comparison of the study arms concerning the primary and secondary end criteria of the study | LSF 2 years after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Dietz, Dr. med., Study Director — University of Leipzig
Locations (27):
- Austria (3):
  - Universitätsklinik für HNO, Graz
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Germany (24):
  - Helios Klinikum Erfurt GmbH Klinik für HNO-Heilkunde, Plastische Operationen, Erfurt, Thuringia
  - Universitätsklinik Aachen, Aachen
  - Charité, Campus Benjamin Franklin, Berlin
  - Klinikum Neukölln, Vivantes GmbH, Berlin
  - Klinikum Bielefeld-Mitte, Bielefeld
  - Universitätsklinik Köln, Cologne
  - Malteser Krankenhaus St. Anna gGmbH, HNO-Klinik, Duisburg
  - Klinikum Fulda gAG, Klinik für Hals-Nasen-Ohrenkrankheiten, Fulda
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Hannover Nordstadt, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - St. Vincentius Kliniken, Karlsruhe
  - Klinikum Kassel GmbH, Kassel
  - Katholisches Klinikum Koblenz Marienhof, Koblenz
  - Universitätsklinikum Leipzig, Leipzig
  - Universtitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum Großhadern, München
  - Medizinische Fakultät der Westfälischen Wilhelms-Universität Münster, Münster
  - Südharz-Krankenhaus Nordhausen gGmbH, Nordhausen
  - Klinikum Ernst von Bergmann gGmbH, Potsdam
  - Universtitätsklinikum Regensburg, Regensburg
  - Klinikum Stuttgart Katharinenhospital, Klinik für HNO-Krankheiten, Stuttgart
  - Bayerischen Julius Maximillians-Universtät Würzburg, Würzburg

REFERENCES:
- [Derived] Dietz A, Wichmann G, Kuhnt T, Pfreundner L, Hagen R, Scheich M, Kolbl O, Hautmann MG, Strutz J, Schreiber F, Bockmuhl U, Schilling V, Feyer P, de Wit M, Maschmeyer G, Jungehulsing M, Schroeder U, Wollenberg B, Sittel C, Munter M, Lenarz T, Klussmann JP, Guntinas-Lichius O, Rudack C, Eich HT, Foerg T, Preyer S, Westhofen M, Welkoborsky HJ, Esser D, Thurnher D, Remmert S, Sudhoff H, Gorner M, Bunzel J, Budach V, Held S, Knodler M, Lordick F, Wiegand S, Vogel K, Boehm A, Flentje M, Keilholz U. Induction chemotherapy (IC) followed by radiotherapy (RT) versus cetuximab plus IC and RT in advanced laryngeal/hypopharyngeal cancer resectable only by total laryngectomy-final results of the larynx organ preservation trial DeLOS-II. Ann Oncol. 2018 Oct 1;29(10):2105-2114. doi: 10.1093/annonc/mdy332. PMID 30412221